CLINICAL TRIAL: NCT06401005
Title: A Single-arm, Open, Phase II Clinical Study of SBRT, Chemotherapy, and Cadonilimab (AK104) Neoadjuvant Therapy for Triple-negative Breast Cancer (TNBC)
Brief Title: SBRT, Chemotherapy, and AK104 Neoadjuvant Therapy for Triple-negative Breast Cancer (TNBC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, professor, Hubei Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBCH-RT-2024-02
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TNBC patients (Experimental)
  Interventions: Drug: Cadonilimab (AK104)

INTERVENTIONS:
Drug: Cadonilimab (AK104) — 8Gy*3 SBRT to irradiate the primary lesion (without axillary lymph node metastasis) or 6Gy*3 SBRT irradiation to irradiate the primary lesion and axillary lymph node metastasis will be administered at first. And then the first cycle of chemotherapy+AK104 given within 24 hours of the end of SBRT. The total eight cycles of preoperative chemotherapy combined with immunotherapy were administered. Surgical resection was performed within 4-6 weeks after the completion of the eighth cycle of chemotherapy combined with immunotherapy. The chemotherapy regimen consisted of: Four cycles of doxorubicin 50mg/m2 (Q3W) + cyclophosphamide 600mg/m2 (Q3W) were administered, followed by four cycles of sequential albumin paclitaxel (125 mg/m2, d1, d8) and carboplatin (AUC=6, d1, Q3W) for 4 cycles. Postoperative completion of 9 cycles of immunotherapy was continued ± the need for postoperative adjuvant radiotherapy was confirmed based on the patient's preoperative status.

SUMMARY:
Studies have indicated that the improvement in pathological complete response (pCR) is significantly correlated with triple-negative breast cancer（TNBC）patients' overall survival (OS). Patients with TNBC have poor efficacy for neoadjuvant chemotherapy. The combination of neoadjuvant therapy with immunotherapy and chemotherapy has been demonstrated to enhance the pCR rate of TNBC patients, increasing it from 45% to approximately 60%. Therefore, how to further improve the pCR rate of TNBC breast cancer became the main objective of this study. Stereotactic radiotherapy (SBRT) not only kills tumor cells directly, but also kills the distant unirradiated tumor cells by promoting the cross-initiation of tumor-specific CD8+ T cells, a phenomenon known as the abscopal effect. Our research team has recently discovered that the triple therapy model of SBRT + anti-vascular targeting + anti-PD-1 was safe and efficacious in lung cancer patients. Cadonilimab (AK104) is an PD-1/CTLA-4 bispecific antibody. In order to improve the pCR, a single-arm, open, phase II clinical study was proposed to explore the safety and efficacy of SBRT+AK104+chemotherapy, a neoadjuvant treatment modality, in the treatment of TNBC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed ER-/PR-/HER2- invasive breast cancer patients (ER/PR immunohistochemistry negative or<1%; Her2 immunohistochemistry of 0, 1+, or 2+/FISH-) patients; patients meeting one of the following conditions: (1) tumor mass larger than 2cm, (2) the presence of axillary lymph node metastasis, and (3) the desire to conserve breasts, but the ratio of tumor size to breast volume is large and difficult to conserve breasts;
2. Patients aged ≥18 years old;
3. ECOG score of 0-1;
4. Biochemical test indexes before enrollment must meet the following criteria, hematologic: white blood cell count (WBC) ≥ 2.0x10^9/L; neutrophil count (ANC) ≥ 1.5×10^9/L; platelet count (PLT) ≥ 100×10^9/L; hemoglobin (Hb) ≥ 90g/L; function: total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN); glutamate aminotransferase (ALT) ≤3 × ULN; aspartate aminotransferase (AST) ≤3 × ULN; renal function: creatinine (Cr) ≤1.5 × ULN; if >1.5 × ULN, creatinine clearance needs to be ≥50mL/min (calculated according to Cockcroft-Gault formula); coagulation: activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 × ULN.

Exclusion Criteria:

1. Received chemotherapy, targeted therapy, or radiation therapy within 12 months prior to first use of study drug;
2. Solid organ or blood system transplantation;
3. Myocardial infarction, poorly controlled arrhythmia (including QTc intervals ≥ 470 ms) within 6 months prior to first use of study drug (QTc intervals are calculated using the Fridericia formula, which is: QTc=QT/RR ^0.33);
4. Class III-IV cardiac insufficiency according to NYHA criteria or cardiac ultrasound: LVEF < 50%;
5. poorly controlled hypertension (defined as systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg), previous hypertensive crisis or hypertensive encephalopathy;
6. Human immunodeficiency virus (HIV) infection, HIV-positive; active tuberculosis; previous and current subjects with interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-associated pneumonitis, and severely impaired lung function that may interfere with the detection and management of suspected drug-associated pulmonary toxicity;
7. Known active or suspected autoimmune disease;
8. Subjects who are allowed to enroll in a stable state and do not require systemic immunosuppressive therapy;
9. Who have received a live vaccine within 28 days prior to the first use of study drug; however, inactivated viral vaccines for seasonal influenza are allowed;
10. Who require systemic treatment with corticosteroids (> 10 mg/day prednisone equivalent dose) or other immunosuppressive medications within 14 days prior to the first use of study drug or for the duration of the study. Subjects. However, enrollment will be permitted in the absence of active autoimmune disease if the subject is treated with topical or inhaled steroids (low potency), systemic short-term use in small doses, single paracortical/intra-articular injections, or adrenocorticotropic hormone replacement therapy at a dose of ≤ 10 mg/day prednisone equivalent; and if any active infections that require systemic administration of Active infection requiring systemic administration of anti-infective therapy; subjects receiving prophylactic antibiotic therapy (e.g., for prevention of urinary tract infections or chronic obstructive pulmonary disease) are eligible for enrollment;
11. Hepatitis B (those with a positive Hepatitis B Surface Antigen [HBsAg] or Hepatitis B Core Antibody [HBcAb] test and positive Hepatitis B Virus Deoxyribonucleic Acid [HBV-DNA] test), Hepatitis C (those with a positive Hepatitis C Virus [HCV] antibody test and positive Hepatitis C Virus [HBV] antibody test), and Hepatitis C (those with a positive Hepatitis B virus [HCV] antibody test and positive Hepatitis C Virus [HCV] antibody test) antibody test positive and hepatitis C virus ribonucleic acid [HCV-RNA] test positive); subjects with hepatitis B and hepatitis C co-infection (positive HBsAg or HBcAb test and positive HCV antibody test);
12. Who have received other antibodies/drugs targeting immune checkpoints in the past, such as anti-PD-1, anti-PD-L1, anti-cytotoxic T-lymphocyte associated antigen- 4 (CTLA-4), and anti-cytotoxic T-lymphocyte associated antigen- 4 (CTLA-4). 4 (CTLA-4), etc.; are participating in another clinical study or are planning to start this study treatment less than 14 days from the end of treatment in the previous clinical study;
13. Have undergone major surgery within 4 weeks prior to the first dose of study drug. Definition of major surgery for this study: surgery that requires at least 3 weeks of postoperative recovery time before receiving treatment on this study. Tumor puncture or lymph node excision biopsy allowed for enrollment;
14. Pregnant or lactating females with a known history of severe allergy to any monoclonal antibody or the study drug and its excipients;
15. Known history of psychotropic substance abuse or drug use; discontinued use of alcohol allowed for enrollment;
16. Subjects with other factors that, in the judgment of the investigator, make them unsuitable for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-11-28 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete pathologic remission (pCR) rate | Up to the 30 weeks
  pCR is defined as ypT0/Tis and ypN0

SECONDARY OUTCOMES:
Objective response rate | Up to the 30 weeks
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.
EFS | Up to 12 months after surgery
  Event free survival
Quality of life assessment | Up to 12 months after surgery
  Using the EORTC QLQ-BR2. It is based on the core cancer scale EORTCQLQ1-C30 with 23 additional scales specific to breast cancer patients. The questions are specified in the QLQ1C30, and by summing all the questions, a score (0-100) is obtained that is positively related to the quality of life of breast cancer patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China